CLINICAL TRIAL: NCT06518018
Title: Exploring the Efficacy and Safety of High-Dose Rate Brachytherapy Combined with Immunotherapy and Chemotherapy As a Second-Line Treatment in Patients with Advanced Non-Small Cell Lung Cancer: a Single-Center, Retrospective, Propensity Score-Matched Study
Brief Title: Efficacy and Safety of High-Dose Rate Brachytherapy with Immunotherapy and Chemotherapy As Second-Line Treatment for Advanced Non-Small Cell Lung Cancer
Acronym: HIBIC-NSCLC
Status: Active, not recruiting | Type: Observational
Sponsor: The First People's Hospital of Neijiang (Other)
Responsible Party: Principal Investigator, Ou Jiang, Chief of Cancer Center, Neijiang No.2 People's Hospital
Other Study IDs: lunshen（yan）2023.no 10
Record Dates: First submitted 2024-07-13; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Advanced Stage NSCLC; Second-line Treatment; Patients Without Targetable Driver Mutations
Keywords: Second-Line Treatment; High-Dose Rate (HDR) Brachytherapy; Non-Small Cell Lung Cancer (NSCLC); Immune Checkpoint Inhibitors (ICIs); Propensity Score-Matched; Advanced Stage
MeSH Terms: conditions — Barakat syndrome; Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Study Group: HDR Brachytherapy + Immunotherapy + Chemotherapy Group
  Interventions: Radiation: HDR brachytherapy (30Gy single fraction)
- Control Group: Immunotherapy + Chemotherapy Group
  Interventions: Drug: Immunotherapy

INTERVENTIONS:
Radiation: HDR brachytherapy (30Gy single fraction) — Study Group receives a novel triple combination therapy for advanced NSCLC in the second-line setting. The treatment begins with a single fraction of high-dose rate (HDR) brachytherapy, delivering 30 Gy locally to the tumor site. This is followed within 1-3 days by systemic therapy, combining immunotherapy and chemotherapy , both administered intravenously.
  Other Names: ICIs; chemotherapy
  Groups: Study Group
Drug: Immunotherapy — Control Group receives the current standard of care for second-line treatment of advanced NSCLC. This regimen consists of a combination of immunotherapy and chemotherapy , both administered intravenously
  Other Names: chemotherapy
  Groups: Control Group

SUMMARY:
This is a single-center, retrospective, propensity score-matched study exploring the efficacy and safety of high-dose rate (HDR) brachytherapy combined with immune checkpoint inhibitors (ICIs) and chemotherapy as a second-line treatment for advanced non-small cell lung cancer (NSCLC).

The study will compare two groups:

Study group: HDR brachytherapy (30Gy single fraction) + ICIs (pembrolizumab) + chemotherapy (docetaxel) Control group: ICIs (pembrolizumab) + chemotherapy (docetaxel) alone Primary objective: To assess the objective response rate (ORR)

Secondary objectives: To evaluate progression-free survival (PFS), overall survival (OS), disease control rate (DCR), and safety.

The study aims to address the unmet clinical need for effective treatments in advanced NSCLC patients who have progressed after immunotherapy. It will investigate whether the addition of HDR brachytherapy to immunotherapy and chemotherapy can improve treatment outcomes.

This research is significant as it explores a novel treatment combination, potentially offering new options for second-line treatment of advanced NSCLC. It also aims to contribute to the understanding of how radiotherapy doses affect immunotherapy responses and may help identify biomarkers for treatment response prediction.

DETAILED DESCRIPTION:
Study Title: Exploring the Efficacy and Safety of High-Dose Rate Brachytherapy Combined with Immunotherapy and Chemotherapy as a Second-Line Treatment in Patients with Advanced Non-Small Cell Lung Cancer

Background:

Non-small cell lung cancer (NSCLC) is a significant health concern in China, accounting for approximately 18.1% of new cancer cases in 2022. Despite advancements in targeted therapies and immunotherapies, patients with advanced NSCLC who progress after initial treatment face limited options and poor prognosis. This study aims to address this unmet clinical need by investigating a novel combination therapy.

Objectives:

Primary: To evaluate the objective response rate (ORR) of high-dose rate (HDR) brachytherapy combined with immune checkpoint inhibitors (ICIs) and chemotherapy in advanced NSCLC patients.

Secondary: To assess progression-free survival (PFS), overall survival (OS), disease control rate (DCR), and safety of the combination therapy.

Study Design:

This is a single-center, retrospective, propensity score-matched study comparing two treatment approaches:

Study group: HDR brachytherapy + ICIs + chemotherapy Control group: ICIs + chemotherapy alone

Treatment Protocol:

Study group: Patients will receive HDR brachytherapy (30Gy single fraction), followed by pembrolizumab and docetaxel chemotherapy within 1-3 days.

Control group: Patients will receive pembrolizumab and docetaxel chemotherapy without brachytherapy.

Key Scientific Questions:

Evaluate the potential improvement in second-line treatment efficacy for advanced NSCLC patients through the combination therapy.

Investigate the mechanisms by which HDR brachytherapy enhances the effectiveness of ICIs and chemotherapy.

Analyze the differential efficacy of the combination therapy across various subgroups of NSCLC patients.

Rationale:

Recent evidence suggests that radiotherapy can exert immunomodulatory effects, potentially enhancing immune treatment responses. High-dose radiotherapy has been shown to improve local control and survival rates in early-stage NSCLC when combined with immunotherapy. This study extends this concept to advanced NSCLC as a second-line treatment option.

Significance:

This research addresses a critical gap in current treatment options for advanced NSCLC patients who have progressed after immunotherapy. It aims to:

Improve patient outcomes in terms of quality of life and survival. Advance scientific understanding of the interaction between radiotherapy and immunotherapy.

Explore potential biomarkers for treatment response prediction. Contribute to the development of more personalized treatment strategies in oncology.

Innovation:

This is the first study to investigate HDR brachytherapy combined with ICIs and chemotherapy for previously treated advanced NSCLC patients. The novel combination strategy shows potential for improved efficacy and safety, offering new options for second-line treatment of advanced NSCLC.

Expected Outcomes:

The study aims to demonstrate improved ORR, PFS, and OS in the combination therapy group compared to the control group. It also seeks to establish the safety profile of the combination therapy and identify patient subgroups that may benefit most from this approach.

Conclusion:

This study represents a significant step towards addressing the unmet needs of advanced NSCLC patients who have progressed after initial treatment. By exploring this innovative combination therapy, the research aims to contribute valuable insights to the field of oncology and potentially improve treatment outcomes for this challenging patient population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced Non-Small Cell Lung Cancer (NSCLC),Likely stage IIIB-IV, though specific staging is not mentioned
* Patients requiring second-line treatment Implying progression after first-line therapy
* Age: Adults (specific age range not provided, but typically 18 years or older)
* Presence of measurable disease according to RECIST v1.1 criteria
* Adequate organ function (specific parameters not provided, but typically included in such studies)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 (not explicitly stated, but common in similar studies)

Exclusion Criteria:

* Presence of targetable driver mutations (e.g., EGFR, ALK, ROS1, BRAF)
* Prior treatment with HDR brachytherapy for the current disease
* Contraindications to immunotherapy or chemotherapy
* Severe comorbidities that would preclude safe administration of study treatments
* Brain metastases, unless treated and stable (not explicitly stated, but common in similar studies)
* Participation in another clinical trial with an investigational agent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Adult patients with advanced Non-Small Cell Lung Cancer (NSCLC)
  2. Requiring second-line treatment after progression on initial therapy
  3. Likely stage IIIB-IV disease
  4. Measurable disease according to RECIST v1.1 criteria
  5. Without targetable driver mutations (e.g., EGFR, ALK, ROS1, BRAF)
  6. Candidates for immunotherapy and chemotherapy
  7. Adequate organ function to tolerate proposed treatments
  8. ECOG performance status likely 0-2
  9. May have prior exposure to immunotherapy
  10. Treated at a single center in China
  11. Divided into two groups
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Every 8 weeks from baseline up to 24 months or until disease progression, unacceptable toxicity, or withdrawal from the study, whichever occurs first
  The proportion of patients achieving either a complete response (CR) or partial response (PR) according to RECIST v1.1 criteria

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Progression-Free Survival was assessed from the date of treatment initiation until the date of first documented disease progression or death from any cause, whichever occurred first, assessed up to 24 months.
  Time from treatment initiation to disease progression or death from any cause

OTHER OUTCOMES:
Overall Survival (OS) | Overall Survival was measured from the date of treatment initiation until death from any cause or patients who were still alive at the last follow-up were censored at that time point, assessed up to 36 months.
  Time from treatment initiation to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- The Second People's Hospital of Neijiang, Neijiang, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will not be shared due to patient privacy concerns, institutional policies, regulatory compliance issues in China, consent limitations in this retrospective study, and the sensitive nature of cancer treatment data. However, the study protocol and statistical analysis plan may be available upon reasonable request to the principal investigator, subject to institutional review board approval and compliance with privacy regulations. Aggregate results and analyses are expected to be published in peer-reviewed journals and presented at scientific conferences. While individual data sharing is not possible, the research team may be open to discussing potential collaborative projects or secondary analyses with interested researchers, subject to necessary approvals and ethical considerations.

REFERENCES:
- [Background] Chen HY, Xu L, Li LF, Liu XX, Gao JX, Bai YR. Inhibiting the CD8+ T cell infiltration in the tumor microenvironment after radiotherapy is an important mechanism of radioresistance. Sci Rep. 2018 Aug 9;8(1):11934. doi: 10.1038/s41598-018-30417-6. PMID 30093664
- [Background] Tateishi Y, Takeda A, Horita N, Tsurugai Y, Eriguchi T, Kibe Y, Sanuki N, Kaneko T. Stereotactic Body Radiation Therapy With a High Maximum Dose Improves Local Control, Cancer-Specific Death, and Overall Survival in Peripheral Early-Stage Non-Small Cell Lung Cancer. Int J Radiat Oncol Biol Phys. 2021 Sep 1;111(1):143-151. doi: 10.1016/j.ijrobp.2021.04.014. Epub 2021 Apr 21. PMID 33891980
- [Background] Weichselbaum RR, Liang H, Deng L, Fu YX. Radiotherapy and immunotherapy: a beneficial liaison? Nat Rev Clin Oncol. 2017 Jun;14(6):365-379. doi: 10.1038/nrclinonc.2016.211. Epub 2017 Jan 17. PMID 28094262
- [Background] Twyman-Saint Victor C, Rech AJ, Maity A, Rengan R, Pauken KE, Stelekati E, Benci JL, Xu B, Dada H, Odorizzi PM, Herati RS, Mansfield KD, Patsch D, Amaravadi RK, Schuchter LM, Ishwaran H, Mick R, Pryma DA, Xu X, Feldman MD, Gangadhar TC, Hahn SM, Wherry EJ, Vonderheide RH, Minn AJ. Radiation and dual checkpoint blockade activate non-redundant immune mechanisms in cancer. Nature. 2015 Apr 16;520(7547):373-7. doi: 10.1038/nature14292. Epub 2015 Mar 9. PMID 25754329
- [Background] Zhang Z, Liu X, Chen D, Yu J. Radiotherapy combined with immunotherapy: the dawn of cancer treatment. Signal Transduct Target Ther. 2022 Jul 29;7(1):258. doi: 10.1038/s41392-022-01102-y. PMID 35906199
- [Background] Wu M, Liu J, Wu S, Liu J, Wu H, Yu J, Meng X. Systemic Immune Activation and Responses of Irradiation to Different Metastatic Sites Combined With Immunotherapy in Advanced Non-Small Cell Lung Cancer. Front Immunol. 2021 Dec 14;12:803247. doi: 10.3389/fimmu.2021.803247. eCollection 2021. PMID 34970277
- [Background] Chen D, Song X, Wang H, Gao Z, Meng W, Chen S, Ma Y, Wang Y, Li K, Yu J, Yue J. Previous Radiotherapy Increases the Efficacy of IL-2 in Malignant Pleural Effusion: Potential Evidence of a Radio-Memory Effect? Front Immunol. 2018 Dec 11;9:2916. doi: 10.3389/fimmu.2018.02916. eCollection 2018. PMID 30619280
- [Background] Ko EC, Raben D, Formenti SC. The Integration of Radiotherapy with Immunotherapy for the Treatment of Non-Small Cell Lung Cancer. Clin Cancer Res. 2018 Dec 1;24(23):5792-5806. doi: 10.1158/1078-0432.CCR-17-3620. Epub 2018 Jun 26. PMID 29945993
- [Background] Shabason JE, Minn AJ. Radiation and Immune Checkpoint Blockade: From Bench to Clinic. Semin Radiat Oncol. 2017 Jul;27(3):289-298. doi: 10.1016/j.semradonc.2017.03.002. Epub 2017 Mar 16. PMID 28577836
- [Background] Taniguchi Y, Shimokawa T, Takiguchi Y, Misumi T, Nakamura Y, Kawashima Y, Furuya N, Shiraishi Y, Harada T, Tanaka H, Miura S, Uchiyama A, Nakahara Y, Tokito T, Naoki K, Bessho A, Goto Y, Seike M, Okamoto H. A Randomized Comparison of Nivolumab versus Nivolumab + Docetaxel for Previously Treated Advanced or Recurrent ICI-Naive Non-Small Cell Lung Cancer: TORG1630. Clin Cancer Res. 2022 Oct 14;28(20):4402-4409. doi: 10.1158/1078-0432.CCR-22-1687. PMID 35980349
- [Background] Gandhi SJ, Minn AJ, Vonderheide RH, Wherry EJ, Hahn SM, Maity A. Awakening the immune system with radiation: Optimal dose and fractionation. Cancer Lett. 2015 Nov 28;368(2):185-90. doi: 10.1016/j.canlet.2015.03.024. Epub 2015 Mar 20. PMID 25799953
- [Background] Garon EB, Hellmann MD, Rizvi NA, Carcereny E, Leighl NB, Ahn MJ, Eder JP, Balmanoukian AS, Aggarwal C, Horn L, Patnaik A, Gubens M, Ramalingam SS, Felip E, Goldman JW, Scalzo C, Jensen E, Kush DA, Hui R. Five-Year Overall Survival for Patients With Advanced Non-Small-Cell Lung Cancer Treated With Pembrolizumab: Results From the Phase I KEYNOTE-001 Study. J Clin Oncol. 2019 Oct 1;37(28):2518-2527. doi: 10.1200/JCO.19.00934. Epub 2019 Jun 2. PMID 31154919
- [Background] Spigel DR, Faivre-Finn C, Gray JE, Vicente D, Planchard D, Paz-Ares L, Vansteenkiste JF, Garassino MC, Hui R, Quantin X, Rimner A, Wu YL, Ozguroglu M, Lee KH, Kato T, de Wit M, Kurata T, Reck M, Cho BC, Senan S, Naidoo J, Mann H, Newton M, Thiyagarajah P, Antonia SJ. Five-Year Survival Outcomes From the PACIFIC Trial: Durvalumab After Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. J Clin Oncol. 2022 Apr 20;40(12):1301-1311. doi: 10.1200/JCO.21.01308. Epub 2022 Feb 2. PMID 35108059
- [Background] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leal TA, Riess JW, Jensen E, Zhao B, Pietanza MC, Brahmer JR. Five-Year Outcomes With Pembrolizumab Versus Chemotherapy for Metastatic Non-Small-Cell Lung Cancer With PD-L1 Tumor Proportion Score >/= 50. J Clin Oncol. 2021 Jul 20;39(21):2339-2349. doi: 10.1200/JCO.21.00174. Epub 2021 Apr 19. PMID 33872070
- [Background] Shi JF, Wang L, Wu N, Li JL, Hui ZG, Liu SM, Yang BY, Gao SG, Ren JS, Huang HY, Zhu J, Liu CC, Fan JH, Zhao SJ, Xing PY, Zhang Y, Li N, Lei WD, Wang DB, Huang YC, Liao XZ, Xing XJ, Du LB, Yang L, Liu YQ, Zhang YZ, Zhang K, Qiao YL, He J, Dai M; LuCCRES Group. Clinical characteristics and medical service utilization of lung cancer in China, 2005-2014: Overall design and results from a multicenter retrospective epidemiologic survey. Lung Cancer. 2019 Feb;128:91-100. doi: 10.1016/j.lungcan.2018.11.031. Epub 2018 Nov 24. PMID 30642458
- [Background] Xia C, Dong X, Li H, Cao M, Sun D, He S, Yang F, Yan X, Zhang S, Li N, Chen W. Cancer statistics in China and United States, 2022: profiles, trends, and determinants. Chin Med J (Engl). 2022 Feb 9;135(5):584-590. doi: 10.1097/CM9.0000000000002108. PMID 35143424